CLINICAL TRIAL: NCT01971931
Title: Prospective Evaluation of Biomarkers Variability in Knee Prosthetic Surgery
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Assistant Professor, University of Milan
Other Study IDs: BioBone01
Record Dates: First submitted 2013-07-05; First posted 2013-10-30 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, tibial bone biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing TKR.

SUMMARY:
Bone quality is an important factor influencing the outcome of total knee replacement (TKR) surgery. Therefore, assessing bone quality preoperatively could help the surgeon in the choice of the most appropriate prosthetic implant.

The primary goal of this study is to measure serum and tissue levels of some proteins involved in bone remodelling.

DETAILED DESCRIPTION:
Aseptic implant loosening after TKR causes knee pain, reduces knee function and may require revision surgery.

Several proteins have been identified, which are involved in bone metabolism and remodelling; variations in serum levels of some of these proteins after TKR loosening have also been described.

However, preoperative identification of risk factors for aseptic loosening remains a challenge.

An observational study is conducted to evaluate how levels of the following serum biomarkers vary after TKR:

* osteoprotegerin (OPG)
* receptor activator of nuclear factor kappa-B (RANK)
* receptor activator of nuclear factor kappa-B ligand (RANK-L)
* sclerostin
* cathepsin K

To avoid bias caused by inflammatory states, C reactive protein (CRP), interleukin 1 (IL-1), interleukin 6 (IL-6), tumor necrosis factor α (TNF-α) levels and erythrocyte sedimentation rate (ESR) will be measured.

Secondary goals are to evaluate the mRNA expression of OPG, RANK-L, cathepsin K and sclerostin on tibial bone biopsies and to study if changes in serum biomarkers levels after surgery are associated with:

* clinical outcomes
* periprosthetic bone density
* variation of two bone reabsorption markers, the postoperative change of which has already been described in details: type 1 collagen cross-linked C-terminal telopeptide (CTP1) and type 1 procollagen N-terminal telopeptide (P1NP).

One day before surgery, after having signed informed consent, patients will undergo a vertebral and femoral dual-energy X-ray absorptiometry (DEXA) scan and blood samples will be collected.

During surgery a tibial biopsy will be collected. Between 4 and 7 days postoperatively and 3, 6 and 12 months after surgery patients will again undergo periprosthetic DEXA scans and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40, <80
* Indication for TKR
* Surgical indication for PFC Sigma®, posterior stabilized, mobile bearing TKR
* Patients signed written informed consent

Exclusion Criteria:

* Age > 80, < 40
* TKR revision surgery
* Fixed knee deformities greater than 15° in varus, valgus, flexion or tibial slope.
* Knee ankylosis
* Paget's disease
* Hyperparathyroidism
* Patient treated with: bisphosphonates, strontium ranelate, selective estrogen receptor modulators for osteoporosis, calcitonin, denosumab.
* Informed consent not accepted
* Serious comorbidity
* Active infections
* Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TKR surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers serum level after surgery | One day before surgery; 3 months after surgery and 12 months after surgery
  OPG, RANK, RANK-L, sclerostin, cathepsin K, CTP1 and P1NP levels will be assessed on blood samples. CRP, IL-1, IL-6, TNF-α and ESR will also be measured to identify inflammatory states.

SECONDARY OUTCOMES:
Change in periprosthetic bone density after surgery | 3, 6, 12 months after surgery
  Variations of tibial bone density will be evaluated repeating DEXA scans 3, 6 and 12 months after surgery. A preoperative vertebral and femoral DEXA scan will be used to estimate patient's initial bone density.
Biomarkers mRNA expression | Baseline
  OPG, RANK-L , cathepsin K, sclerostin and CTP1 mRNA levels will be estimated using Real-Time polymerase chain reaction (RT-PCR) on tibial plateau biopsies. RT-PCR will be performed simultaneously on all samples, after collection of all biopsies.

OTHER OUTCOMES:
Change in knee function score after surgery | One day before surgery; 3, 6, 12 months after surgery
  For evaluation of knee function, patients will be asked to fill in the Oxford Knee Score (OKS) questionnaire.
Change in knee pain scale after surgery | One day before surgery; 3, 6, 12 months after surgery
  For evaluation of knee pain, patients will be asked to indicate their knee pain on a visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Galliera, PhD, Principal Investigator — Istituto Ortopedico Galeazzi IRCCS, Milano, Italy; Randelli Pietro, MD, Study Director — Policlinico San Donato IRCCS, San Donato Milanese, Italy; Corsi Romanelli M. Massimiliano, MD, Principal Investigator — Policlinico San Donato IRCCS, San Donato Milanese, Italy
Locations (1):
- Policlinico San Donato (Istituto di Ricovero e Cura a Carattere Scientifico), San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vega D, Maalouf NM, Sakhaee K. CLINICAL Review #: the role of receptor activator of nuclear factor-kappaB (RANK)/RANK ligand/osteoprotegerin: clinical implications. J Clin Endocrinol Metab. 2007 Dec;92(12):4514-21. doi: 10.1210/jc.2007-0646. Epub 2007 Sep 25. PMID 17895323
- [Background] Colombini A, Lombardi G, Galliera E, Dogliotti G, Randelli P, Meerssemann A, Mineo G, Cabitza P, Corsi MM. Plasma and drainage fluid levels of soluble receptor activator of nuclear factor-kB (sRANK), soluble receptor activator of nuclear factor-kB ligand (sRANKL) and osteoprotegerin (OPG) during proximal humerus fracture healing. Int Orthop. 2011 May;35(5):777-82. doi: 10.1007/s00264-010-1088-3. Epub 2010 Jul 11. PMID 20623281
- [Background] Rogers A, Eastell R. Circulating osteoprotegerin and receptor activator for nuclear factor kappaB ligand: clinical utility in metabolic bone disease assessment. J Clin Endocrinol Metab. 2005 Nov;90(11):6323-31. doi: 10.1210/jc.2005-0794. Epub 2005 Aug 16. PMID 16105967
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Li MG, Thorsen K, Nilsson KG. Increased bone turnover as reflected by biochemical markers in patients with potentially unstable fixation of the tibial component. Arch Orthop Trauma Surg. 2004 Jul;124(6):404-9. doi: 10.1007/s00402-004-0695-0. Epub 2004 May 20. PMID 15156331
- [Background] Li MG, Nilsson KG. The effect of the preoperative bone quality on the fixation of the tibial component in total knee arthroplasty. J Arthroplasty. 2000 Sep;15(6):744-53. doi: 10.1054/arth.2000.6617. PMID 11021450
- [Background] Mertens MT, Singh JA. Biomarkers in arthroplasty: a systematic review. Open Orthop J. 2011 Mar 16;5:92-105. doi: 10.2174/1874325001105010092. PMID 21584201
- [Background] Kenanidis EI, Potoupnis ME, Papavasillioul KA, Sayegh FE, Petsatodis GE, Kapetanos GA. Serum levels of bone turnover markers following total joint arthroplasty. J Orthop Surg (Hong Kong). 2010 Dec;18(3):290-5. doi: 10.1177/230949901001800307. PMID 21187538
- [Background] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091
- [Background] van Loon CJ, Oyen WJ, de Waal Malefijt MC, Verdonschot N. Distal femoral bone mineral density after total knee arthroplasty: a comparison with general bone mineral density. Arch Orthop Trauma Surg. 2001 May;121(5):282-5. doi: 10.1007/s004020000232. PMID 11409560
- [Background] Minoda Y, Ikebuchi M, Kobayashi A, Iwaki H, Inori F, Nakamura H. A cemented mobile-bearing total knee replacement prevents periprosthetic loss of bone mineral density around the femoral component: a matched cohort study. J Bone Joint Surg Br. 2010 Jun;92(6):794-8. doi: 10.1302/0301-620X.92B6.23159. PMID 20513875
- [Background] Soininvaara TA, Harju KA, Miettinen HJ, Kroger HP. Periprosthetic bone mineral density changes after unicondylar knee arthroplasty. Knee. 2013 Mar;20(2):120-7. doi: 10.1016/j.knee.2012.10.004. Epub 2012 Nov 13. PMID 23154036
- [Derived] Cucchi D, Menon A, Galliera E, Messina C, Zanini B, Marazzi MG, Massaccesi L, Compagnoni R, Corsi Romanelli MM, Randelli P. A Prospective Assessment of Periprosthetic Bone Mineral Density and Osteoimmunological Biomarkers Variations After Total Knee Replacement Surgery. J Clin Densitom. 2019 Jan-Mar;22(1):86-95. doi: 10.1016/j.jocd.2018.05.039. Epub 2018 May 26. PMID 30072203